CLINICAL TRIAL: NCT03780517
Title: A Phase 1 Study of BOS172738 in Patients With Advanced Solid Tumors With RET Gene Alterations Including Non-Small Cell Lung Cancer (NSCLC) and Medullary Thyroid Cancer (MTC)
Brief Title: Safety, Efficacy, and Tolerability of BOS172738 in Patients With Advanced Rearranged During Transfection (RET) Gene-Altered Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BOS172738-01; 2018-002612-27 (EudraCT Number)
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Advanced Nonhaematologic Malignancies
Keywords: BOS172738; RET gene; Medullary Thyroid Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 2a; Carcinoma, Medullary; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BOS172738 (Experimental): In Part A (dose escalation), participants with advanced solid tumors with rearranged during transfection (RET) gene alterations will receive oral BOS172738 at a starting dose of 10 milligrams (mg) once daily in each 28-day cycle. In Part B (dose expansion), participants with RET gene-fusion non-small cell lung cancer (NSCLC), with RET gene-mutant medullary thyroid cancer (MTC), and with RET gene-altered advanced tumors or NSCLC/MTC with prior specific RET gene-targeted therapy will be enrolled in Cohorts 1, 2, and 3, respectively, and will receive oral BOS172738 once daily in each 28-day cycle at the recommended Phase 2 dose (RP2D) established in Part A.
  Interventions: Drug: BOS172738

INTERVENTIONS:
Drug: BOS172738 — Oral capsules

SUMMARY:
This study will be conducted to assess the safety and tolerability of BOS172738 when administered to patients with advanced solid tumors with rearranged during transfection (RET) gene alterations and also to establish the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of BOS172738.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Male or female participants must be ≥ 18 years, at the time of signing the informed consent
* Diagnosis of advanced solid tumor with a documented rearranged during transfection (RET) gene altered malignancy as determined locally by a DNA based assay of tumor tissue and/or blood
* Participants must have no alternative approved therapy.
* For participants in Part B expansion cohort only: documented local diagnosis of either 1) advanced RET gene fusion non-small cell lung cancer (NSCLC); 2) advanced RET gene mutant medullary thyroid cancer (MTC); or 3) other RET gene altered advanced tumors or NSCLC/MTC with prior specific RET gene targeted therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Negative pregnancy test for females of child bearing potential; must be surgically sterile, postmenopausal, or willing and able to be compliant with a contraceptive regimen
* Contraceptive use by men or women should be consistent with local regulations.
* Capable of giving signed informed consent

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Inability to take oral medications or gastrointestinal (GI) conditions that can interfere with the swallowing or absorption of study medication
* Uncontrolled or severe concurrent medical condition
* History of upper GI bleeding, ulceration, or perforation within 12 months prior to the first dose of study drug
* Known history of stroke or cerebrovascular accident within 6 months prior to the first dose of study drug
* Participants with known infection with human immunodeficiency virus (HIV) or Acquired Immune Deficiency Syndrome (AIDS) (testing not required)
* Participants who are hepatitis B surface antigen positive or participants who are hepatitis C antibody positive (Participants who have been successfully treated for hepatitis C virus [HCV] are eligible if an undetectable HCV viral load at least 6 months after completion of treatment can be demonstrated.)
* Any evidence of serious active infections
* Uncontrolled or severe cardiovascular disease
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements
* Participants with a prior or concurrent malignancy other than the malignancies under study
* Ongoing cancer directed therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with any treatment-emergent (TE) serious adverse event (SAE) | a minimum of approximately 3 months
Number of participants with any non-serious TEAE | a minimum of approximately 3 months
Number of participants with grade 3, grade 4, or grade 5 TEAEs | a minimum of approximately 3 months
Number of participants with any related TEAE | a minimum of approximately 3 months
Number of participants with any TEAE leading to study drug discontinuation | a minimum of approximately 3 months
Maximum tolerated dose (MTD) of BOS172738 | throughout Cycle 1 (each cycle is 28 days)
Recommended phase 2 dose (RP2D) of BOS172738 | 28-day cycles in Part A (minimum of one dose of BOS172738 received)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | a minimum of approximately 3 months
Objective Disease Control Rate (ODCR) | a minimum of approximately 3 months
Progression-Free Survival (PFS) | a minimum of approximately 3 months
Duration of Response (DoR) | a minimum of approximately 3 months
Time to Response (TTR) | a minimum of approximately 3 months
Duration of Complete Response (DoCR) | a minimum of approximately 3 months
Part A: Plasma concentration of BOS172738 | Pre-dose on Days 1, 2, 15, and 16 of Cycle 1; Day 1 of Cycles 2, 3, and 4. 15 minutes (min); 30 min; 1, 3, 6, 8, 10, and 12 hours after the BOS1722722 dose on Days 1 and 15 of Cycle 1 (each cycle is 28 days)
Part B: Plasma concentration of BOS172738 | Pre-dose on Day 1 of Cycles 2, 3, and 4 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (2):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - UZ Leuven, Leuven
- France (4):
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - Hôpital Pitié-Salpêtrière, Paris
  - Institut Gustave Roussy, Villejuif
- Prince of Wales Hospital, Hong Kong, Hong Kong
- South Korea (5):
  - Chungbuk National University Hospital, Cheongju-si
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Seoul
- Spain (5):
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Germans Trias i Pujol, Badalona
  - Instituto Oncológico Dr. Rosell, S.L., Barcelona
  - Start Madrid - Ciocc, Madrid
  - START MADRID-FJD, Hospital Fundación Jiménez Díaz, Madrid
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei